CLINICAL TRIAL: NCT05299957
Title: Usefulness of Integrated PET/MRI in Oropharyngeal Squamous Cell Carcinoma Evaluation
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ng, Shu-Hang, Professor, Chang Gung Memorial Hospital
Other Study IDs: 201407314A3
Record Dates: First submitted 2022-03-07; First posted 2022-03-29 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Oropharyngeal Cancer
Keywords: Oropharyngeal cancer; integrated PET/MR
MeSH Terms: conditions — Oropharyngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- oropharyngeal squamous cell carcinoma: a total of 160 patients with histologically proven oropharyngeal SCC subjected to chemoradiation will be enrolled. Exclusion criteria include previous head or neck malignant tumor, a second malignant tumor, distant metastasis, contraindications to MRI (renal insufficiency, cochlear implant, cardiac pacemaker, or intracranial aneurysmal ferromagnetic clips), and serum glucose level >200 mg/dl. Each enrolled patients will undergo detail clinical examination, including human papillomavirus test.
  Interventions: Diagnostic Test: PETMRI

INTERVENTIONS:
Diagnostic Test: PETMRI — PET/MRI data will be acquired on the integrated PET/MRI scanner. After fast-view T1-weighted MR localizer sequence for scout imaging and Dixon VIBE sequence for attenuation correction, a whole-body PET scan will be performed to cover from the head to the proximal thigh, with an acquisition time of 4 min per bed position. Simultaneously, whole body MR image acquisition will be performed with the axial HASTE sequence and coronal STIR sequence as well as the sagittal T1-weighted Turbo spine echo and STIR sequence. Afterwards, regional PET and MRI images will be simultaneously performed. DWI will be performed using a single shot spin-echo echo-planar technique. A total of 10 b values will be used for the reconstruction of IVIM and kurtosis imaging. DCE-PWI will be acquired by using a 3D T1-weighted spoiled gradient-echo sequence. Thereafter, dedicated regional MRI will be obtained. Finally, whole body axial VIBE with fat saturation will be performed.

SUMMARY:
Head and neck cancer (HNC) continues to be a significant health care problem in Taiwan and oropharyngeal squamous cell carcinoma (SCC) is the common subtype. With the concern of organ preservation in recent years, concurrent chemoradiation is the major treatment modality for oropharyngeal SCC, while endoscopy with biopsy serves as the main diagnostic tools. With the advance of MRI technology, whole body MRI is now possible, and functional techniques become more feasible in the head and neck region, including diffusion-weighted imaging (DWI) which comprises of monoexponential DWI, intravoxel incoherent motion (IVIM) model and Kurtosis (biexponential or non-Gaussian fitting), and dynamic contrast-enhanced perfusion weighted MRI (DCE-PWI) become feasible. Therefore, MRI can evaluate distant site status of HNC in the single examination session and provide biologic information of tumors. Positron emission tomography/CT (PET/CT) is another common imaging modality to evaluate HNC, because of its ability to provide whole-body anatomic and metabolic information.

Integrated PET/MRI is a novel imaging technology that combines PET and MRI in one single scanner. In this 3-year prospective study, the investigators will take the advantages of integrated PET/MRI scanner with DWI (including monoexponential, kurtosis and IVIM modes) and DCE-PWI to evaluate our 160 patients with oropharyngeal SCC subjected to chemoradiation. Non-contrast chest CT will also be performed on the same day. The investigators aim to determine whole-body staging/restaging accurately, to predict treatment response and prognosis, and to determine necessity of noncontrast chest CT. The investigators expect that this project will offer the validation of usefulness of integrated PET/MRI in tumor staging/restaging of oropharyngeal SCC and resultant clinical impact. The role of noncontrast chest CT in the workup with our PET/MRI protocol can be defined. It will also provide evidence about how and to what extent the various simultaneously acquired MRI and PET functional parameters can help prediction of treatment response and prognosis of oropharyngeal SCC subjected to chemoradiation, which are important in timely modification of treatment regimen.

DETAILED DESCRIPTION:
In this three-year prospective project, a total of 160 patients with histologically proven oropharyngeal SCC subjected to chemoradiation will be enrolled. Exclusion criteria include previous head or neck malignant tumor, a second malignant tumor, distant metastasis, contraindications to MRI (renal insufficiency, cochlear implant, cardiac pacemaker, or intracranial aneurysmal ferromagnetic clips), and serum glucose level >200 mg/dl. Each enrolled patients will undergo detail clinical examination, including human papillomavirus test. The participants will undergo low dose chest CT on the same day before PET/MRI. In the posttreatment period, baseline whole body MRI will be obtained 3 months after chemoradiation. Thereafter, the participants will then be followed up also with alternative extend-field CT and whole body MRI by every 6 months. If tumor recurrenceis confirmed or highly suspected, PET/MRI will also be performed for tumor re-staging.

The three-years planning Adequate cases number and follow-up duration are essential for statistical analysis and outcome determination of oropharyngeal SCC treated with chemoradiation. The investigators plan to accomplish this study in 3 years.

In the first year, the works of the this project in the first year will design the data bank categories, set up the workflow and optimize the imaging protocols, determine the diagnostic capability of MRI component, PET component, integrated PET/MRI in tumor staging, determinate any added diagnostic value of noncontrast chest CT in integrated PET/MRI, and study the early treatment response and the patterns of residual tumor.

In the second year, the investigators will continue to the first-year works, and further include the following works to determinate incidence and predictors of treatment failure of oropharyngeal SCC, and to study the patterns of treatment response and early recurrence. In the third year, the investigators will continue to do previous work and will also get sufficient sample size to perform statistical analysis of the relationship between the imaging parameters and patient outcomes, attain comprehensive imaging about patterns of tumor recurrence and posttreatment changes/complications, investigate to what extent biologic imaging parameters may affect outcome and patient selection for chemoradiation, and analysis the accuracy, pitfalls and cost effectiveness of the PET/MRI alone and PET/MRI with noncontrast chest CT in evaluating in patients with oropharyngeal SCC.

PET/MRI data will be acquired on the integrated PET/MRI scanner , which acquires simultaneous PET and MR data with a 3.0-T magnet. The examination protocol will combined a whole-body scan with a dedicated examination of the head and neck area. All participants will fast for 6 h before the scan. At 50-70 min post injection of 370 MBq of FDG, the patient will be placed on the PET/MRI scanner bed. After fast-view T1-weighted MR localizer sequence for scout imaging and Dixon VIBE sequence for attenuation correction, a whole-body PET scan will be performed in 5 bed positions to cover from the head to the proximal thigh, with an acquisition time of 4 min per bed position. Simultaneously, whole body MR image acquisition will be performed for the corresponding 5 bed positions with the axial HASTE sequence and coronal STIR sequence as well as the sagittal T1-weighted Turbo spine echo(TSE) and STIR sequence.

Afterwards, regional PET and MRI images will be simultaneously performed. Regional PET will be performed with an acquisition time of 10 min, while a dedicated MRI of the head and neck region will be acquired in the axial and coronal projections with T1-weighted TSE sequence and T2-weighted TSE sequence with fat saturation. Axial DWI will be performed using a single shot spin-echo echo-planar technique with modified Stejskal-Tanner diffusion gradient pulsing scheme. A total of 10 b values will be used for the reconstruction of IVIM and kurtosis imaging, which are: 0, 20, 40, 80, 100, 200, 400, 800, 1200, 1500 sec/mm2. DCE-PWI at the head and neck region will be acquired by using a 3D T1-weighted spoiled gradient-echo sequence. A spatial saturation slab will be implanted inferior to the acquired region to minimize the inflow effect from the carotid arteries. Before the contrast agent administration, baseline longitudinal relaxation time values will be calculated from image acquired with different flip angles. Then, the dynamic series will be acquired using the same sequence with a 15° flip angle, after intravenous administration of paramagnetic contrast agent at 3 ml/s. Thereafter, dedicated regional MRI will be obtained with T1-weighted TSE sequence with fat saturation in the axial and coronal projections. Finally, whole body axial VIBE with fat saturation will be performed. The total acquisition time is about 42 min, and the mean in-room time for PET/MR will be approximately 60 min.

Non-enhanced low-dose chest CT Spiral low-dose chest CT without contrast material enhancement will be performed before PET/MRI on the same examination day. Acquisition parameters include peak voltage of 120 kVp, mAs of 50, collimation of 64x0.5 mm and reconstruction interval of 3-mm.

Data analysis Readers are aware that patients have oropharyngeal SCC, and they will be blinded to the results of other studies and to PET/MR data. The PET, MRI and chest CT images will be first interpreted independently. All images will be then reviewed together and compared. A checklist of various distributions of tumor extension, nodal spread and distant metastasis will be recorded. The clinical and imaging findings will be discussed jointly by the Head-and-Neck research team. Endoscopic biopsy, ultrasonographic guided fine needle aspiration or CT-guided biopsy will be performed in any lesions suspicion for malignancy if possible. If biopsy of the lesion of interest is not feasible, or yields a negative result, close clinical and imaging follow-up will be pursued. All participants will be followed up for at least 12 months. The clinical and functional imaging data will be collected and analyzed for predicting treatment response and prognosis. For the diffusion MRI, regions of interest will be manually placed on the lesions on ADC map to encompass as much of the solid tumor area as possible. The signal intensities measured on the images acquired at different b-values S(b) will be numerically fitted against the model, S(b)=S0 e-b*ADC, where S0 and Sb are signal intensities at different b values, For IVIM imaging, the relationship between signal intensities and b values can be expressed by the equation: Sb/S0 = (1-f )．exp(-bD) + f．exp[-b( D + D＊)] where f is a microvascular volume fraction representing the fraction of the diffusion linked to microcirculation, D represents pure diffusion coefficient, and D* is perfusion-related incoherent microcirculation. For the DKI, the relationship between signal intensities and b values can be expressed by the equation: ln[S(b)] = ln[S(0)] - b x Dapp + 1/6b2 x Dapp2 x Kapp where S is the signal intensity (arbitrary units), b is the b-value (s/mm2), Dapp is the apparent diffusion coefficient (10-3 mm2/s), and Kapp is the apparent kurtosis coefficient denoting thedeviation from a Gaussian distribution. We will also perform monoexponential fitting by using Kapp=0 in the equation, yielding ADCmono. For the DCE-PWI MRI, the change in contrast agent concentration over time, Ct(t), will be determined in each voxel in the tumor, and the compartmental tracer kinetic model will be applied to each voxel by using an arterial input function, Cp(t), measured in each individual: Ct (t)=VpCp(t) + Ktrans ∫0 t Cp(t' ) exp(Ktrans(t-t') /Ve )dt' where t' is the time (in minutes) as an integration variable, and Cp(t') is the concentration of contrast agent in the blood plasma as a function of time.

For PET imaging parameters, SUV and MTV of the target lesions will be measured from attenuation-corrected 18F-FDG PET images by drawing the boundaries drawn large enough to include the lesions. An SUV threshold of 2.5 will be used to delineate the MTV. The TLG is calculated as the product of the mean SUV and the MTV.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven oropharyngeal SCC subjected to chemoradiation

Exclusion Criteria:

* previous head or neck malignant tumor, a second malignant tumor, distant metastasis, contraindications to MRI (renal insufficiency, cochlear implant, cardiac pacemaker

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in a tertiary referral center
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Primary tumor staging of oropharyngeal cancer by PET/MR | 2 years
  correlation of size of primary tumor(cm), size of metastatic nodes (cm), and number of distant metastasis with PET, MRI and PET/MR

SECONDARY OUTCOMES:
Survival of oropharyngeal cancer by FDG uptake of PETMT | 4 years
  correlate survival rates with SUV, Ktrans(min-1), Kep(min-1), Ve, ADC (mm2/s)

CONTACTS AND LOCATIONS:
Overall Officials: WU SHU-CHIEN, Principal Investigator — Department of Medic Imaging and Intervention, Chang Gung Memorial Hospital
Locations (1):
- Department of Medical Imaging and Intervention, Chang Gung Memorial Hospital, Guishan, Taoyuan, Taiwan